CLINICAL TRIAL: NCT06772740
Title: Randomized Clinical Trial of Middle Meningeal Artery Embolization for Patients With Chronic Subdural Hematoma (COMPLEMENT Study)
Brief Title: Middle Meningeal Artery Embolization for Patients With Chronic Subdural Hematoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kazutaka Uchida (Other)
Responsible Party: Sponsor-Investigator, Kazutaka Uchida, Associate Professor (Stroke Center), Hyogo Medical University
Organization: Hyogo Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R000063204
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Endovascular Treatment; Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatments with middle meningeal artery embolization (Experimental)
  Interventions: Procedure: Middle meningeal artery embolization
- Conventional treatments alone (No Intervention)

INTERVENTIONS:
Procedure: Middle meningeal artery embolization — Middle meningeal artery embolization within 7 days after randomization
  Arms: Conventional treatments with middle meningeal artery embolization

SUMMARY:
COMPLEMENT study (ChrOnic subdural hematoMa Patients suppLemented with Embolization of Middle mENingeal artery Trial) is a prospective, open label, blinded endpoint (PROBE), Japanese, two-arm, randomized, controlled, post-market study to assess the efficacy and safety of middle meningeal artery embolization for chronic subdural hematoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18
2. pre-mRS 0-3
3. Hematoma thickness >=10mm
4. Having at least one risk factor Risk factor: Age >=75, Antithrombotic therapy, DM, Bilateral hematoma, Markwalder grading score >3, Preoperative volume >=130ml, Preoperative midline shift >=8mm, CT appearance (Homogeneous, laminar or separated)

Exclusion Criteria:

1. Cr >=1.8
2. Plt <50,000, PT-INR >2
3. Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence of chronic subdural hematoma | 6 months after randomization
  Recurrence of chronic subdural hematoma is defined as the maximum thickness of subdural hematoma exceeding 10 mm or the patient receiving re-operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hyogo Medical University, Nishinomiya, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No